CLINICAL TRIAL: NCT02890927
Title: Quasi-experimental Before-and-after Study to Compare the Effectiveness of Geriatric Co-management on Preventing Functional Decline as Compared to Standard of Care in Older Cardiology Patients
Brief Title: Geriatric-CO-mAnagement for Cardiology Patients in the Hospital
Acronym: G-COACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 22/15/028
Record Dates: First submitted 2016-08-24; First posted 2016-09-07 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Geriatric Assessment; Health Services for the Aged; Cardiovascular Diseases; Activities of Daily Living; Delirium; Frail Elderly; Length of Stay
Keywords: Geriatric Nursing; Geriatric co-management; Geriatric team
MeSH Terms: conditions — Cardiovascular Diseases; Delirium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cardio-geriatric co-management (Experimental): A geriatric co-management intervention will be implemented on the cardiology units of the University Hospitals Leuven. Geriatric co-management is defined as a shared responsibility and decision making between the cardiology team and the geriatric team who provides complementary medical care in the prevention and management of geriatric problems. Patients included in the co-management program will undergo a comprehensive geriatric assessment within 24 hours of hospital admission.
  Interventions: Other: Cardio-geriatric co-management
- Standard of care (No Intervention): The control group will receive the standard of care on the cardiology units. This includes multidisciplinary care with a one weekly multidisciplinary team meeting. Team members include a cardiology resident (supervised by a cardiologist), ward nurses, a physical therapist, a social worker and a dietician. A geriatric consultation team is available for consultation services if requested by the cardiology team.

INTERVENTIONS:
Other: Cardio-geriatric co-management — A comprehensive geriatric assessment on admission will stratify patients in groups:
  1. Low risk patients are expected to do well and will not receive co-management.
  2. Medium risk patients are expected to develop complications. A geriatric nurse will visit the cardiology wards daily to co-manage these patients aiming to prevent complications by coordinating interdisciplinary care, implementing protocols, perform assessments and bedside education. The geriatric nurse will work collaboratively with the cardiology ward staff based on a shared decision making. Patients will receive early rehabilitation and discharge planning.
  3. High risk patients have an acute geriatric syndrome. The geriatric nurse will visit the cardiology wards (see above), and a geriatrician will co-manage the acute geriatric syndrome(s). The geriatrician will work collaboratively with the cardiology ward staff based on a shared decision making. Patients will receive early rehabilitation and discharge planning.
  Arms: Cardio-geriatric co-management

SUMMARY:
The primary objective of the evaluation study is to determine if geriatric co-management is superior to standard of care in preventing functional decline in older patients admitted for acute heart disease or Transcatheter Aortic Valve Implementation (TAVI) to the cardiology units of the University Hospitals Leuven.

DETAILED DESCRIPTION:
This study aims to implement and evaluate a geriatric co-management intervention in older patients admitted for acute heart disease or Transcatheter Aortic Valve Implementation (TAVI) to the cardiology units of the University Hospitals Leuven. The study uses a mixed-methods methodology aiming to 1) assess the feasibility and evaluate the effectiveness of geriatric co-management, 2) describe the experiences of intervention participants, and 3) perform a process evaluation. We will first consecutively recruit patients on the cardiology units to measure the standard of care in the control group. The geriatric co-management intervention will then be implemented and piloted on the participating units. Once fully implemented, we will consecutively recruit patients for the intervention group who will receive the geriatric co-management intervention.

ELIGIBILITY:
Inclusion Criteria: Patients will be included if they:

* Are admitted for non-surgical treatment of an acute heart problem (patients may be admitted through the emergency department or the cardiology outpatient services for any heart related acute disease) OR if they are admitted for Transcatheter Aortic Valve Implantation (TAVI);
* Are aged 75 years or older;
* Have an expected length of stay of three days or longer;
* Non-palliative on hospital admission
* Are Dutch speaking and testable;
* Give informed consent or proxy-informed consent;

Exclusion Criteria: Patients will be excluded if they:

* Are admitted from another hospital unit or other hospital;
* Have been admitted to the intensive care unit for three days or longer;

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 454 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Functional status on activities of daily living assessed using the Katz Index of Activities of Daily Living. | Hospital admission (baseline) up to hospital discharge around an average of 12 days.
  A difference of 1 point on the Katz Index will be considered clinically relevant.
Functional decline in activities of daily living assessed using the Katz Index of Activities of Daily Living | Hospital admission (baseline) up to hospital discharge around an average of 12 days.
  A decline of 1 point between admission and discharge on the Katz Index will be considered clinically relevant.

SECONDARY OUTCOMES:
Functional decline in activities of daily living assessed using the Barthel Index of Activities of daily. Living. | Hospital admission (baseline), hospital discharge around an average of 12 days, and at 30 days, 3 months and 6 months follow-up after hospital discharge.
Community mobility assessed using the Life-Space assessment. | Hospital admission (baseline), and at 30 days, 3 months and 6 months follow-up after hospital discharge.
Short Physical Performance Test (SPPB). | Hospital admission (baseline), up to at hospital discharge around an average of 12 days.
  The SPPB consist of gait speed, balance test, and chair stand test.
Peak handgrip force assessed at the dominant side with the elbow at 90° of flexion, and the forearm and wrist in a neutral position. | Hospital admission (baseline) up to hospital discharge around an average of 12 days.
  Isometric handgrip force will be measured with a hydraulic hand dynamometer (Jamar dynamometer; JA Preston Corporation; Jackson, MI).
Symptomatic infections defined by a clinical diagnosis of pneumonia, urinary tract infection, sepsis and wound infection. | Hospital admission (baseline) up to hospital discharge around an average of 12 days.
Delirium assessed using the 3D confusion assessment method. | Hospital admission (baseline) and on day 3, 5, 7 and 9 (or every day when a patient is delirious).
Cognitive status assessed using the Mini-Cog. | Hospital admission (baseline) up to hospital discharge around an average of 12 days.
Falls and fall related injuries. | Hospital admission (baseline), hospital discharge around an average of 12 days, and at 30 days, 3 months and 6 months follow-up after hospital discharge.
  A fall incident is defined as an unexpected event in which the patient comes to rest on the ground, floor or lower level. Fall related injuries will be divided in two groups: minor and major.
Obstipation assessed using nurses recorded observations. | Hospital admission (baseline) up to hospital discharge around an average of 12 days.
  Obstipation is defined as not having passed stool in five days or more.
Length of hospital stay. | Hospital admission (baseline) up to hospital discharge around an average of 12 days.
Institutionalization. | hospital discharge around an average of 12 days, and at 30 days, 3 months and 6 months follow-up after hospital discharge.
  New admission to nursing home or skilled nursing facility
Thirty day unplanned readmission rate. | 30 days follow-up after hospital discharge.
Survival | Hospital discharge around an average of 12 days, and at 30 days, 3 months and 6 months follow-up after hospital discharge.
  Time to death
Quality of life assessed using the EQ-5D. | Hospital admission (baseline), hospital discharge around an average of 12 days, and at 30 days, 3 months and 6 months follow-up after hospital discharge.
Quality of life index assessed by converting the EQ-5D using standardized index values. | Hospital admission (baseline), hospital discharge around an average of 12 days, and at 30 days, 3 months and 6 months follow-up after hospital discharge.
Functional status on activities of daily living assessed using the Katz Index of Activities of Daily Living. | At 30 days, 3 months and 6 months follow-up after hospital discharge.
  Functional status will be measured using the Katz Index of Activities of Daily Living.
Unplanned hospital readmissions | up to 6 months follow-up after hospital discharge
  Time to the first unplanned hospital readmission
Hospital costs | Between hospital admission and discharge, an average of 12 days
  Costs registered for to the treatment, care, logistics and stay in the hospital

OTHER OUTCOMES:
Experiences by the intervention participants using focus group discussions and individual interviews. | Through study completion, an average of 1 year.
  The interviews will focus on implementation determinants and the interaction of the intervention with the context in which it was implemented.
Reach of the intervention using structured observations and process indicators. | Through study completion, an average of 1 year.
  Reach is defined as the number of eligible patients receiving the intervention.
Fidelity of the intervention using structured observations and process indicators. | Through study completion, an average of 1 year.
  Fidelity is defined as the extent to which the intervention was implemented as defined in the protocol.
Dose of the intervention using structured observations and process indicators. | Through study completion, an average of 1 year.
  Dose is defined as the number of intervention components delivered as defined in the protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Flamaing, PhD, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Koen Milisen, PhD, MSN, Principal Investigator — University of Leuven; Mieke Deschodt, PhD, MSN, Principal Investigator — University of Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Deschodt M, Van Grootven B, Jeuris A, Devriendt E, Dierckx de Casterle B, Dubois C, Fagard K, Herregods MC, Hornikx M, Meuris B, Rex S, Tournoy J, Milisen K, Flamaing J. Geriatric CO-mAnagement for Cardiology patients in the Hospital (G-COACH): study protocol of a prospective before-after effectiveness-implementation study. BMJ Open. 2018 Oct 21;8(10):e023593. doi: 10.1136/bmjopen-2018-023593. PMID 30344179